CLINICAL TRIAL: NCT05517408
Title: Dose Exploration of Ciprofol for Sedation in Gastrointestinal Endoscopic Diagnosis and Treatment of Obese Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: diansansu0722
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Gastric Cancer; Gastric Ulcer; Intestinal Polyps; Intestinal Cancer
Keywords: sedation; gastrointestinal endoscopy; obese patient; ciprofol
MeSH Terms: conditions — Stomach Neoplasms; Stomach Ulcer; Intestinal Polyps; Intestinal Neoplasms | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ciprofol group (Experimental)
  Interventions: Drug: ciprofol

INTERVENTIONS:
Drug: ciprofol — The first patient received Ciprofol 0.3mg/kg (actual body weight) at a rate of 1 mg/s. If the desired depth of sedation/anesthesia reached, then it was judged as negative, and the dose of Ciprofol in next patient would be decreased by one concentration gradient (the difference between two adjacent drugs was 1:1.1); If the desired sedation/anesthesia depth was not achieved, then it was judged as positive. And the dose of Ciprofol in next patient would be increased by one concentration gradient. Patients were enrolled consecutively until the trial was terminated at the eighth crossing point (positive to negative or negative to positive).

SUMMARY:
Ciprofol is a new anesthetic, which combines with γ- Aminobutyric acid-a (GABAA) receptor. Ciprofol has shown equivalent anesthetic efficacy of propofol at 1/4 to 1/5 of the dosage. Ciprofol has the pharmacodynamic characteristics of rapid onset, stable and rapid recovery. Phase III clinical results showed that the incidence of injection pain and respiratory and circulatory depression of ciprofol was lower than that of propofol. Therefore, ciprofol has a good application prospect in sedation for gastrointestinal endoscopy, especially for obese patients. In the current study, we would explore the proper dose of Ciprofol in sedated gastrointestinal endoscopy in obese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age, ≤18 and ≤60 years, no gender limit
2. Undergoing routine gastrointestinal endoscopic diagnosis and treatment
3. American Society of Anesthesiologists (ASA) classification I-II
4. Body Mass Index(BMI) ≥28kg/m^2
5. Clearly understand and voluntarily participate in the study; provide signed informed consent

Exclusion Criteria:

1. Unhealthy alcohol drinking, defined by more than three standard drinks per day (≈10 g alcohol , equivalent to 50 g of strong Chinese spirits)
2. Drug abuse history within 3 months before the screening period
3. People who are known to be allergic to eggs, bean products, opioids and other drugs, propofol, etc
4. The researcher believes that patients should not participate in this trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2023-08-13 (Estimated)

PRIMARY OUTCOMES:
Calculating the the median effective dose (ED50) of ciprofol for sedation gastrointestinal endoscopy in obese patients. | Patients will be followed for the duration of hospital stay, an expected average of 2 hours

SECONDARY OUTCOMES:
Calculating the the ED95 of ciprofol for sedation gastrointestinal endoscopy in obese patients. | Patients will be followed for the duration of hospital stay, an expected average of 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
We have no plan to share individual participant data.